CLINICAL TRIAL: NCT07295613
Title: Multicenter Prospective Registry of Patients With Hypertrophic Cardiomyopathy
Brief Title: ReGistry of hypeRtrophic cArDIomyopathy: Regional fEatures, geNeTics and Course
Acronym: GRADIENT
Status: Enrolling by invitation | Type: Observational
Sponsor: Central State Medical Academy (Other)
Collaborators: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Principal Investigator, Zateyshchikov Dmitry, MD, PhD, head of the department of therapy, cardiology and functional diagnostic, Central State Medical Academy
Other Study IDs: CGMA 4/1/2023
Record Dates: First submitted 2025-04-13; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hypertrophic Cardiomyopathy (HCM)
Keywords: genetic; epidemiology; Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood samples for subsequent DNA extraction and genetic analysis can be collected at any time of the day, regardless of food intake. Venous blood is collected from the cubital vein in sterile vacutainer tubes with EDTA reagent (purple caps). It is optimal to use 3 4.5 ml tubes. The tubes should be labeled with the patient&#39;s last name and initials, individual code at the participating center, collection date, and sample type (A, B, or C). After blood collection, the tubes should be frozen at an optimal temperature of (-) 200C. The blood is not centrifuged.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is envisioned as the very first of its kind in the Russian Federation, aiming to provide a comprehensive characterization of the clinical spectrum and disease burden, focusing on the epidemiology and progression of HCM in the largest cohort of adult and pediatric patients from this region. This registry will help increase knowledge of the epidemiology and prevalence of HCM, ultimately improving diagnosis and management. To assess the feasibility of new interventions, understanding the epidemiological profile of patients with HCM is essential. Clinical characteristics, imaging patterns, and outcomes may vary across different geographic regions. Completing this registry will enhance our understanding of the disease in Russia, and promote measures that modify the natural history of HCM

DETAILED DESCRIPTION:
This study is observational registry of patients with HCM in Russian Federation. The study seeks to elucidate disease progression, identify contributing clinical factors, and explore new as well as previously established associations between genetic and acquired determinants and clinical features of HCM.The Additional Objectives of the Study are:

* To evaluate the natural progression of HCM in non-operated patients who have indications for myectomy and in high-risk patients for SCD, who have not been implanted with an ICD.
* To clarify the relationship between pediatric and adult HCM by constructing large pedigrees, including clinically and genetically examined relatives.
* To evaluate real-world clinical practices, both surgical and therapeutic, in the management of LV obstruction.
* To investigate the impact of comorbidities on phenotypic expression of HCM.
* To establish a group of national HCM experts and centers of excellence. We plan to include 1400 patients with HCM in the study.The examination of patients includes the collection of clinical information, ECG, EchoCG, Holter ECG monitoring, etc.• During follow-up period, patients or their relatives will be contacted by phone at least once every 12 months
* At follow-up visits, information regarding the study endpoints, ant medical examinations, and interventions that have occurred since the time of enrollment will be collected. Investigators are encouraged to make every effort to obtain official medical records that document these endpoints and any interventions that have taken place.

The genetic study aims to identify the causative genetic variants associated with HCM in enrolled patients (probands). The genetic testing will be conducted using new-generation sequencing (NGS) with target gene panels. In the study cohort of patients, an analysis of the effect of common genetic variants, identified based on the literature or GWAS, on the course of HCM will be conducted. In the study cohort (partially or entirely), genome-wide sequencing might be performed to replicate the significance of existing variants and to identify new genetic determinants that define the development of the HCM phenotype.

A comparative analysis of different parameters will be performed across various subgroups, categorized by the following characteristics (but not limited to them):

* Sex
* Age at first diagnosis
* Proband or relative status
* Presence of LV obstruction
* Morphological type of HCM
* Presence of comorbidities
* Presence of mutations or VUSs in sarcomere genes

In addition to the clinical and genetic spectrum and endpoints, the rate and type of diagnostic and treatment procedures related to HCM will be assessed.

In cases where the diagnosis of HCM was reconsidered or declined based on the results of additional investigations after enrollment, such patients will not be included in the prognosis analysis. However, they will be described in the clinical and genetic profile of the study population.

ELIGIBILITY:
Inclusion Criteria:

* Any age
* Signed informed consent form (ICF) for participation in the study, including genetic testing
* Meets the criteria for HCM HCM Criteria for Probands ≥ 18 Years Based on ECHO or CMR
* End-diastolic LV wall thickness ≥ 15mm in any segment of the LV HCM Criteria for Probands ≥ 18 Years with Arterial Hypertension
* 1st degree of AH: The same ECHO/CMR criteria as patients without AH
* 2nd and 3rd degrees of AH:
* Asymmetric LV hypertrophy: the ratio of septum / LV PW ≥ 1.5 or apical HCM
* If asymmetry < 1.5, the wall thickness must be ≥ 20mm
* For all patients with arterial hypertension, the presence of at least one of the following ECG changes is obligatory:
* Pathological "dagger" Q wave
* T-wave inversion ≥ 3mm in ≥ 2 adjacent leads
* Poor R progression / QS / RV1 > RV2 < RV3 in V1-V4

HCM Criteria for First-degree Relatives ≥ 18 Years Based on ECHO or CMR and ECG:

* End-diastolic LV wall thickness ≥ 13mm in any segment and/or ECG changes in the absence of CAD, such as (at least one of the following):
* Quantitative signs of LV hypertrophy* + repolarization changes
* T wave inversions in at least 2 adjacent leads: ≥ 3mm in V3-V6, I, aVL or ≥ 5mm in II, III, aVF
* Pathological Q waves (> 25% of R) in at least 2 adjacent leads: II, III, aVF (in the absence of left anterior hemiblock) or V1-V4, or I, aVL, V5-V6

  *Presence at least one of the following:
* Sokolow-Lyon index (S in V1 + R in V5 or V6) > 35mm
* R or S in limb leads ≥ 20mm
* S in V1 or V2 ≥ 30mm
* R in V5 or V6 ≥ 30mm HCM Criteria for Children and Adolescents < 18 Years
* End-diastolic LV wall thickness in any segment > 2.5 standard deviations (> 2.5 z-score) above the norms for the index gender, age and weight (or body surface area) in asymptomatic children/adolescents without a family history of HCM
* End-diastolic LV wall thickness in any segment > 2.0 standard deviations (> 2.0 z-score) above the norms for the index gender, age and weight (or body surface area) in children/adolescents with a family history of HCM or a positive genetic test

Exclusion Criteria:

* Uncontrolled arterial hypertension of 2nd - 3rd degree with mild/moderate (< 20mm) or symmetric LV hypertrophy or a "normal" ECG
* Hemodynamically significant congenital or acquired valve heart disease
* Established diagnosis of metabolic, infiltrative, endocrine, or other diseases known as "phenocopies of HCM"

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adult and pediatric patients with HCM
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 3 years
  death from any cause

SECONDARY OUTCOMES:
nonfatal events | 3 years
  1. Appropriate and non-appropriate ICD shocks
  2. Successful resuscitation
  3. Progression of dyspnea to class III/IV according by NYHA
  4. A reduction in LV EF to less than 50%
  5. Hospitalization due to HF requiring parenteral diuretics and/or inotropic therapy
  6. LVAD implantation
  7. Heart transplantation or being on the waiting list
  8. Septal reduction therapy
  9. Non-fatal ischemic strokes
  10. New onset AF
  11. New onset non-sustained VT
  12. New onset Sustained VT
  13. New onset syncope (highly likely arrhythmogenic)
  14. Other non-fatal CV events, including but not limited to MI and pulmonary embolism.

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Central State Medical Academy, Moscow, Moscow Reg
  - CGMA, Moscow

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT07295613/Prot_SAP_000.pdf
  • Informed Consent Form: v4 (2025-12-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT07295613/ICF_001.pdf